CLINICAL TRIAL: NCT00170170
Title: Clinical Predictors of Late-onset CMV Disease in Solid Organ Transplant Recipients: A Strategy to Improve the Benefits and Reduce the Risks of Anti-CMV Prophylaxis
Brief Title: Risk Factors for Cytomegalovirus Disease in Solid Organ Transplantation
Status: Completed | Type: Observational
Sponsor: Mayo Clinic (Other)
Collaborators: Roche Pharma AG (Industry)
Other Study IDs: 2275-04; VAL101
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2010-02-02 (Estimated); Status verified 2010-02

CONDITIONS: Transplantation; Infection; Cytomegalovirus Infections
Keywords: cytomegalovirus
MeSH Terms: conditions — Infections; Cytomegalovirus Infections

STUDY DESIGN:
Time Perspective: Retrospective

SUMMARY:
This study will investigate the clinical variables that may be used to predict who among the solid organ transplant recipients will develop cytomegalovirus (CMV) disease after completing antiviral prophylaxis.

DETAILED DESCRIPTION:
This study will investigate the clinical and laboratory variables that may be used to predict who among the solid organ transplant recipients will develop CMV disease after completing antiviral prophylaxis. This is a retrospective study of patients seen at the Mayo Clinic during the past five years.

ELIGIBILITY:
Inclusion Criteria:

* Recipients of liver, kidney, pancreas, heart or lung transplantation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Recipients of liver, kidney, pancreas, heart or lung transplantation
Sampling Method: Non-Probability Sample
Enrollment: 500 (Actual)
Dates: Start 2004-11; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymund R. Razonable, M.D., Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States